CLINICAL TRIAL: NCT04352205
Title: A Phase 2 Evaluation of Daratumumab-Based Treatment in Newly Diagnosed Multiple Myeloma Patients With Renal Insufficiency
Brief Title: Daratumumab-Based Therapy for the Treatment of Newly Diagnosed Multiple Myeloma With Kidney Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, R. Donald Harvey, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000007; NCI-2020-01133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP4949-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Plasma Cell Myeloma; Renal Failure
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (daratumumab-based treatment) (Experimental): Patients receive daratumumab IV weekly of cycles 1-3 and on day 1 only of cycle 4, bortezomib SC on days 1, 4, 8, and 11, and dexamethasone IV or PO on days 1-4 of cycle 1 and on day 1 of cycles 2-4 and PO on days 8 and 15 of all cycles. Beginning cycle 2, patients may also receive lenalidomide PO daily on days 1-14 or thalidomide PO QD on days 1-21. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Thalidomide

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO and IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Thalidomide — Given PO
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Softenon; Synovir; Talimol; Thalomid

SUMMARY:
This phase II trial studies how well daratumumab-based therapy works in treating patients with newly diagnosed multiple myeloma with kidney failure. Daratumumab-based therapy includes daratumumab, bortezomib, dexamethasone, and thalidomide or lenalidomide. Daratumumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Bortezomib is a drug that prevents myeloma cells from getting rid of their waste products, leading to being targeted for death. Dexamethasone is a steroid that is commonly used, either alone or in combination with other drugs, to treat multiple myeloma. Lenalidomide and thalidomide may stop the growth of multiple myeloma by blocking the growth of new blood vessels necessary for tumor growth. Giving daratumumab, bortezomib, dexamethasone, and thalidomide or lenalidomide may be a good way to treat patients with newly diagnosed multiple myeloma with kidney failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of patients with newly diagnosed myeloma and acute kidney injury (AKI) who have renal function recovery following 2 cycles (6 weeks) of treatment with a daratumumab-based induction regimen.

SECONDARY OBJECTIVES:

I. Overall response rate at the end of 2 and 4 cycles of therapy. II. Adverse event profile of the combination in patients with AKI. III. Pharmacokinetic parameters of maximum concentration (Cmax), area under the curve (AUC), time to maximum concentration (tmax), clearance, and half life (t1/2) of daratumumab in combination treatment in the AKI population.

IV. Global assessment of renal function at cycle initiation including creatinine clearance (CrCl).

V. Timeline of changes in pharmacodynamic markers of light chains, urine paraprotein, and serum paraprotein measures.

OUTLINE:

Patients receive daratumumab intravenously (IV) weekly of cycles 1-3 and on day 1 only of cycle 4, bortezomib subcutaneously (SC) on days 1, 4, 8, and 11, and dexamethasone IV or orally (PO) on days 1-4 of cycle 1 and on day 1 of cycles 2-4 and PO on days 8 and 15 of all cycles. Beginning cycle 2, patients may also receive lenalidomide PO daily on days 1-14 or thalidomide PO once daily (QD) on days 1-21. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Creatinine clearance < 30 mL/min by Cockcroft-Gault (C-G), 24 hour urine collection or the Modification of Diet in Renal Disease (MDRD) methods. The same method used for inclusion will be used for renal response assessment
* Documented multiple myeloma as defined by the International Myeloma Working Group (IMWG) 2014 criteria including: Clonal bone marrow plasma cells >= 10%. In addition, the patient must meet one of the criteria in day (d)1 or d2:

  * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically (one or more of the following):

    * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal (ULN) or > 2.75 mmol/L (>11 mg/dL)
    * Renal insufficiency: creatinine clearance (CrCl) < 30 mL/min
    * Anemia: hemoglobin value of > 2 g/dL below the lower limit of normal, or a hemoglobin value < 10 g/L
    * Bone lesions: 1 or more osteolytic lesions on skeletal radiography, computed tomography (CT), or magnetic resonance imaging (MRI)
* Measurable disease as defined by any of the following:

  * Serum M-protein level >= 1.0 g/dL or urine M-protein level >= 200 mg/24 hours.
  * IgA, IgD, IgE, or IgM multiple myeloma: serum M-protein level >= 0.5 g/dL or urine M-protein level >= 200 mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the urine: serum Ig free light chain (FLC) >= 10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio
* Prior treatment to stabilize the patient with steroids up to 160 mg IV equivalents of dexamethasone is allowed
* Prior treatment to stabilize the patient with bortezomib up to 2 doses of 1.3 mg/m^2 is allowed
* Subject agrees to refrain from blood donations during therapy on study and for 8 weeks after therapy is completed
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Are not planning to donate eggs during the period of study and up to 3 months after the last dose of study drug
  * Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting study drugs
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) and
  * Agree to no sperm donation during the period of study and up to 3 months after the last dose of study drug

Exclusion Criteria:

* Diagnosed with smoldering multiple myeloma (MM), monoclonal gammopathy of undetermined significance, Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, amyloidosis or primary or secondary plasma cell leukemia
* Participant has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination within 21 days before initiation of protocol therapy
* Plasmapheresis within 28 days
* Platelet count =< 75,000 cells/mm^3 at time of screening evaluation. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Participants with an absolute neutrophil count (ANC) =< 1000 cells/mm^3 at time of screening evaluation. Growth factors may not be used to meet ANC eligibility criteria within 14 days of obtaining screening evaluation
* Participants with hemoglobin level < 7.0 g/dL, at time of screening. Transfusion may be used to meet eligibility criteria within 7 days of obtaining screening evaluation
* Participants with hepatic impairment, defined as bilirubin >= 1.5 x institutional upper limit of normal (ULN) or aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]), or alkaline phosphatase >= 3 x institutional ULN, within 21 days of initiation of protocol therapy
* Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg p.o. once daily [q.d.] or its equivalent) for symptom management and comorbid conditions. Doses of corticosteroid should be stable for at least 7 days prior to study treatment.)
* Steroids160 mg IV equivalents of dexamethasone or bortezomib > 2 doses of 1.3 mg/m^2.
* Known significant cardiac abnormalities including:

  * Congestive heart failure, New York Heart Association (NYHA) class III or IV
  * Uncontrolled angina, arrhythmia or hypertension
  * Myocardial infarction within the past six months
  * Any other uncontrolled or severe cardiovascular condition
  * Prior cerebrovascular event with residual neurologic deficit
* Known history of chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal
* Has known history of moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Serious, intercurrent illness including, but not limited to, clinically relevant active infection, uncontrolled diabetes mellitus, or serious co-morbid medical conditions such as chronic restrictive pulmonary disease, and cirrhosis
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as a viremia at least 12 weeks after completion of antiviral therapy)
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are allowed if they have undergone complete resection
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Known severe intolerance to steroid therapy
* Participants with known central nervous system (CNS) involvement
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to dexamethasone, boron or mannitol
* Female participants pregnant or breast-feeding
* Participants who have undergone major surgery =< 4 weeks prior to starting study drug or who have not recovered from side effects of the surgery
* Participants with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
* Prior exposure to anti-CD38 therapy
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of study medications
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Change in creatinine clearance | Screening until end of Cycle 4 at day 1(12 weeks), each cycle=21 days
  Renal function comparisons of creatinine clearance between methods for the cohort will be conducted, with the primary objective of change from baseline, using the same formula, serving as the analysis dataset.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of Cmax | Cycle 1 at day 1 (12 weeks) to Cycle 2 at Day 15 (12 Weeks), each cycle=21 days
  Maximum concentrations for each patient obtained at the end of daratumumab infusion.
Pharmacokinetic parameters of AUC | Starting at Cycle 1 at day 1(12 weeks) to Cycle 2 at Day 15 (12 weeks), each cycle=21 days
  Area under the plasma concentration time curve from time 0-24 hours and extrapolated to infinity to understand dose exposures.
Pharmacokinetic parameters of CI | Cycle 1 at day (12 weeks) 1 to Cycle 2 at Day 15 (12 weeks), each cycle=21 days
  Clearance for each patient to assess the effect of renal insufficiency and potential changes with myeloma treatment that includes daratumumab.
Incidence of adverse events | Through study completion, an average of 1 year
  Will track grade 3, 4, and 5 adverse events collected clinically in the routine course of care, with particular interest in those associated with daratumumab. Subject incidence of all treatment emergent adverse events of interest will be tabulated by system organ class and preferred term. Tables of fatal adverse events, serious adverse events, adverse events leading to withdrawal from investigational product, other protocol-required therapies or from study, and adverse events of interest will also be provided. Relevant laboratory and vital sign (temperature, heart rate, respiratory rate, and blood pressure) data will be displayed by visit and time (when available), with Common Terminology Criteria for Adverse Events (CTCAE). Additionally, all laboratory data will be summarized by CTCAE grade, again, with grade 3, 4 and 5 values to be collected.
Overall response rate | Through study completion, an average of 1 year
  All efficacy assessments will follow International Myeloma Working Group (IMWG) uniform response criteria and be performed every cycle. Will be defined as the proportion of best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR).
Best overall response | Through study completion, an average of 1 year
  All efficacy assessments will follow IMWG uniform response criteria and be performed every cycle.
Progression free survival | Time from randomization date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Will be defined as number of months from subject's first study dose date to the earlier of disease progression or death due to any cause.
Duration of response | Time from initiation of first response to first documented progression or death, from any cause, whichever came first, assessed up to 100 months
  Will be summarized for all subjects overall, by formulation, by dose cohort level, and by formulation and dose cohort level along with 95% confidence intervals when applicable. Duration of therapy, dose density, and frequency of dose holds or reductions will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: R. Donald Harvey, PharmD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.